CLINICAL TRIAL: NCT06731543
Title: Development of a Condition Specific Quality of Life Scale for Atrial Fibrillation: AF-PROMS
Brief Title: Development of an AF Specific Quality of Life Questionnaire: AF-PROMS
Acronym: AF-PROMS
Status: Active, not recruiting | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: City, University of London (Other)
Responsible Party: Principal Investigator, Prof Richard Schilling, Professor Richard Schilling, Barts & The London NHS Trust
Other Study IDs: Version 5. 14/July/2014
Record Dates: First submitted 2015-09-14; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

GROUPS / COHORTS (1):
- Patients who have atrial fibrillation
  Interventions: Other: No interventions will be made

INTERVENTIONS:
Other: No interventions will be made

SUMMARY:
This study is aiming to develop a Health Related Quality of Life (HRQoL) scale for patients who have atrial fibrillation (AF).

DETAILED DESCRIPTION:
This study is aiming to develop and validate a Health Related Quality of Life (HRQoL) scale for patients who have atrial fibrillation (AF). As this questionnaire is currently under development, it is anticipated this measure will be a short questionnaire which will measure various aspects of quality of life. Once the questionnaire has been validated further details of the final metric used and aspects of quality of life covered in the questionnaire can be provided.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrial fibrillation (AF)

Exclusion Criteria:

* Exclude any participants who it is felt participation will cause distress.
* Exclude participants who do not give consent to take part in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with atrial fibrillation (AF)
Sampling Method: Non-Probability Sample
Enrollment: 206 (Estimated)
Dates: Start 2014-02-14 (Actual); Primary Completion 2026-09-09 (Estimated); Study Completion 2026-09-09 (Estimated)

PRIMARY OUTCOMES:
No primary outcomes will be measured | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Health NHS Trust, London, United Kingdom